CLINICAL TRIAL: NCT07109557
Title: The Effect of Baduanjin on Pain, Comfort, and Quality of Recovery in Patients Undergoing Knee Replacement Surgery
Brief Title: The Effect of Baduanjin on Patients Undergoing Knee Replacement Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Niran Çoban (Other)
Responsible Party: Sponsor-Investigator, Niran Çoban, Asst.Prof., University of Yalova
Organization: University of Yalova (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NCBN
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Pain, Postoperative; Surgery; Knee Replacement; Nurse's Role
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin (Experimental): Participants in this arm will receive supervised Baduanjin exercises in addition to routine postoperative care. The Baduanjin protocol will begin on Postoperative Day 1 and continue for 3 weeks, with daily practice under guidance. Data collection will be performed at four time points using the Visual Analog Scale (VAS), the General Comfort Questionnaire, and the Quality of Recovery-40 (QoR-40).
  Interview and Application Schedule:
  Interview I (Preoperative): Face-to-face interview one day before surgery; informed consent and sociodemographic data collection
  Interview II (Postoperative Day 1): Start of Baduanjin; baseline assessment with VAS, QoR-40, and Comfort Questionnaire
  Interview III (Postoperative Week 4): Follow-up assessment with VAS, QoR-40, and Comfort Questionnaire
  Interview IV (Postoperative Week 8): Final assessment with VAS, QoR-40, and Comfort Questionnaire
  Interventions: Other: Baduanjin
- Standard care (No Intervention): Description:
  Participants in this arm will receive standard postoperative nursing care and physical therapy, without any complementary intervention. Data will be collected at the same four time points as in the intervention group for comparison purposes.
  Interview and Application Schedule:
  Interview I (Preoperative): Face-to-face interview one day before surgery; informed consent and sociodemographic data collection
  Interview II (Postoperative Day 1): Baseline assessment with VAS, QoR-40, and Comfort Questionnaire
  Interview III (Postoperative Week 4): Follow-up assessment with VAS, QoR-40, and Comfort Questionnaire
  Interview IV (Postoperative Week 8): Final assessment with VAS, QoR-40, and Comfort Questionnaire

INTERVENTIONS:
Other: Baduanjin — Baduanjin exercise
  Arms: Baduanjin

SUMMARY:
This randomized controlled trial aims to evaluate the effects of Baduanjin, a traditional Chinese mind-body exercise, on pain, comfort, and quality of recovery in patients undergoing total knee arthroplasty (TKA). The study will be conducted between July 2025 and July 2026 at Yalova Training and Research Hospital's Orthopedics Clinic. Sixty patients will be randomly assigned into two groups: an intervention group practicing Baduanjin and a control group receiving standard postoperative care. The intervention will begin on the first postoperative day and continue for three weeks. Outcome measures include the Visual Analog Scale (VAS) for pain, the General Comfort Questionnaire, and the Quality of Recovery-40 (QoR-40) questionnaire. These assessments will be conducted weekly for three weeks. The control group will follow routine postoperative care without Baduanjin. The primary objective is to determine whether Baduanjin can improve postoperative outcomes in terms of pain reduction, increased comfort, and better recovery quality.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is one of the most frequently performed orthopedic surgeries, especially among elderly individuals, to relieve pain, improve joint function, and enhance quality of life in patients with advanced knee osteoarthritis. However, the postoperative period can be challenging due to significant pain, reduced comfort, limited mobility, and psychological distress, all of which may negatively affect the recovery process. Effective postoperative management is essential to reduce pain, improve comfort, and enhance the quality of recovery.

Pharmacological treatments are commonly used for postoperative pain management; however, their side effects and limitations have increased interest in complementary and integrative practices. One such practice is Baduanjin, a traditional Chinese mind-body exercise that consists of eight gentle, coordinated movements. These movements integrate physical posture, breathing control, and mental focus to promote physical and emotional well-being. Baduanjin can be practiced while standing or sitting, making it suitable for patients in the postoperative period. Studies suggest that Baduanjin may reduce pain, improve psychological states such as anxiety and depression, and promote faster physical recovery through improved circulation, joint flexibility, and relaxation.

This randomized controlled trial aims to evaluate the effects of Baduanjin exercises on pain intensity, comfort level, and quality of recovery in patients who have undergone total knee arthroplasty. The study will be conducted between July 2025 and July 2026 at Yalova Training and Research Hospital, Orthopedics Clinic. A total of 60 participants will be randomly assigned into two groups using a random number table: a Baduanjin group (intervention) and a control group. The intervention group will perform supervised Baduanjin exercises starting from the first postoperative day for a duration of three weeks. Exercises will be practiced under nurse supervision and consist of the eight classical Baduanjin movements.

Pain, comfort, and quality of recovery will be evaluated at the end of each week using the Visual Analog Scale (VAS), the General Comfort Questionnaire, and the Quality of Recovery-40 (QoR-40) instrument. The control group will receive only routine postoperative care, including standard physical therapy and pain management, and will complete the same assessments at the same time intervals.

The primary hypothesis is that Baduanjin practice will significantly reduce pain, increase comfort levels, and improve the quality of recovery in patients undergoing TKA compared to standard care. The secondary objective is to contribute to the growing body of evidence supporting non-pharmacological, mind-body interventions in postoperative nursing care. Given its accessibility, safety, and ease of learning, Baduanjin may serve as a valuable complementary method to enhance surgical recovery and patient well-being

ELIGIBILITY:
Inclusion Criteria:

* Having undergone Knee Replacement Surgery under general anesthesia

  • 18 years old and over,
* Are in stable condition after surgery,
* Are conscious, and
* Volunteer to participate in the study.

Exclusion Criteria:

* Patients with contraindications to Baduanjin exercises,

  -• Over 70 years old,

  • Using anxiolytic and sedative drugs,
* Patients with any mental illness and those who do not meet the inclusion criteria will not be included in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The Effect of Baduanjin on Pain | 12 month
  Visual Analogue Scale:The Visual Analog Scale is a one-dimensional scale commonly used to measure pain intensity. VAS is a measuring tool with a length of 0-10 cm (0-100 mm).Since the aim of the study is to determine the effect of the non-pharmacological method used on existing pain, VAS will be used in the pain assessment before and after the application.
  (Postoperative Day 1): Baseline assessment with VAS, (Postoperative Week 4): Follow-up assessment with VAS (Postoperative Week 8): Final assessment with VAS
The Effect of Baduanjin on Quality of Recovery | 12 month
  Quality of Recovery-40 (QoR-40): The QoR-40 scale evaluates post-surgical recovery and includes five sub-dimensions: emotional state, physical comfort, patient support, physical independence, and pain. It consists of 40 items, each rated on a 5-point Likert scale (1-5). Subscale scores are calculated by summing relevant items; total scores range from 40 to 200. Higher scores reflect better physical and emotional recovery, while lower scores indicate impaired well-being. The QoR-40 will be administered after transfer to the clinic, before the Su Jok therapy, to assess recovery quality in the first 24 hours post-surgery. Reassessments will be conducted at three time points: (1) Postoperative Day 1 (baseline), (2) Postoperative Week 4 (follow-up), and (3) Postoperative Week 8 (final). This structured approach will provide insight into the patient's recovery progress over time.
The Effect of Baduanjin on Comfort | 12 month
  General Comfort Scale: Developed by Kolcaba, the General Comfort Scale assesses individuals' comfort needs and the effectiveness of nursing interventions. It is structured on a taxonomy with three levels and four dimensions, reflecting the theoretical components of comfort. The scale includes 48 items rated on a four-point Likert scale. Items are a mix of positive and negative statements. In positive items, a score of 4 indicates high comfort, while 1 indicates low comfort. Negative items are reverse-scored before summing. The total score ranges from 48 to 192, with higher scores indicating greater overall comfort. In this study, the scale will be administered at three time points: (1) Postoperative Day 1 (baseline), (2) Postoperative Week 4 (follow-up), and (3) Postoperative Week 8 (final) to evaluate the progression of comfort throughout the recovery process.

CONTACTS AND LOCATIONS:
Overall Officials: NİRAN ÇOBAN, Study Director — https://akademik.yok.gov.tr/AkademikArama/view/viewAuthor.jsp
Locations (1):
- Niran Çoban, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghandali E, Moghadam ST, Hadian MR, Olyaei G, Jalaie S, Sajjadi E. The effect of Tai Chi exercises on postural stability and control in older patients with knee osteoarthritis. J Bodyw Mov Ther. 2017 Jul;21(3):594-598. doi: 10.1016/j.jbmt.2016.09.001. Epub 2016 Sep 10. PMID 28750970
- [Background] Tao T, Shi MP, Tan BY, Zhang XS, Sun FL, Liu BR, Li SJ, Li ZH. Evaluation of traditional Chinese exercise for knee osteoarthritis (KOA): an overview of systematic reviews. Syst Rev. 2024 Jul 18;13(1):187. doi: 10.1186/s13643-024-02606-0. PMID 39026375
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Background] Karaman S, Arici S, Dogru S, Karaman T, Tapar H, Kaya Z, Suren M, Gurler Balta M. Validation of the Turkish version of the Quality of Recovery-40 questionnaire. Health Qual Life Outcomes. 2014 Jan 15;12:8. doi: 10.1186/1477-7525-12-8. PMID 24428925
- [Background] Wang, X., Pi, Y., Chen, B., et al. (2020). Effectiveness of Baduanjin exercise for limb function, activities of daily living, and quality of life in post-stroke patients: A systematic review and meta-analysis. Frontiers in Aging Neuroscience, 12, 123
- [Background] Xiong X, Wang P, Li S, Zhang Y, Li X. Effect of Baduanjin exercise for hypertension: a systematic review and meta-analysis of randomized controlled trials. Maturitas. 2015 Apr;80(4):370-8. doi: 10.1016/j.maturitas.2015.01.002. Epub 2015 Jan 9. PMID 25636242
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748